CLINICAL TRIAL: NCT01969851
Title: A MULTI-CENTER, OPEN-LABEL, EXPLORATORY STUDY TO INVESTIGATE THE SAFETY AND EFFICACY OF LACOSAMIDE AS ADJUNCTIVE THERAPY IN SUBJECTS ≥1 MONTH TO <18 YEARS WITH EPILEPSY SYNDROMES ASSOCIATED WITH GENERALIZED SEIZURES.
Brief Title: A Study to Investigate the Safety and Efficacy of Lacosamide Added to the Patients Current Therapy in Patients Aged 1 Month to Less Than 18 Years Old With Epilepsy Syndromes Associated With Generalized Seizures.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP0966; 2012-001446-18 (EudraCT Number)
Expanded Access: NCT03559673 (No longer available)
Record Dates: First submitted 2013-10-21; First posted 2013-10-25 (Estimated); Results first posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Epilepsy
Keywords: Lacosamide; Vimpat; Epilepsy; Children
MeSH Terms: conditions — Epilepsy | interventions — Lacosamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lacosamide (Experimental)
  Interventions: Drug: Lacosamide

INTERVENTIONS:
Drug: Lacosamide — Oral intake twice daily of tablet (100 mg or 50 mg) or syrup formulation (10 mg/ml).
  Total daily dose will be titrated over a period of 6 weeks with starting dose of 100 mg/day or 2 mg/kg/day up to doses not exceeding 600 mg/day or 12 mg/kg/day tablet or syrup, respectively. Followed by a 12 week maintenance period with stable dosing of at least 200 mg/day or 4 mg/kg/day tablet or syrup, respectively.
  Other Names: Vimpat

SUMMARY:
SP0966 is an exploratory study to investigate safety and efficacy of Lacosamide (LCM) in children with epilepsy syndromes associated with generalized seizures. LCM will be added to current antiepileptic treatment.

DETAILED DESCRIPTION:
SP0966 is a Phase 2, multicenter, open-label exploratory study designed to assess the safety and preliminary efficacy of oral lacosamide as adjunctive therapy for epilepsy syndromes associated with generalized seizures in pediatric subjects ≥1 month to <18 years of age.

ELIGIBILITY:
Inclusion Criteria:

* A signed informed consent has been obtained from the parent/legal representative and assent has been obtained from the subject (when possible)
* Subject and caregiver are willing and able to comply with all study requirements including maintaining a daily seizure diary
* Subject is male or female, ≥1 month to <18 years of age
* Subject has a diagnosis of uncontrolled epilepsy with generalized seizures (Type II) according to the International Classification of Epileptic Seizures (1981). The underlying epilepsy syndrome should be documented. Diagnosis should have been established by clinical history and an Electroencephalogram (EEG) with generalized spike-wave discharges. Documentation of the EEG finding of generalized spike waves (EEG recording or a report) is required. The EEG should have been performed no more than 18 months prior to Visit 1 (with no change to diagnosis or seizure types during this time)
* Subject must have experienced 2 or more events (typical generalized seizures associated with diagnosed epilepsy syndrome) within the 6-week prospective Baseline Period
* Subject is on a stable dosage regimen of 1 to 3 antiepileptic drugs (AEDs). The daily dosage regimen of concomitant AED therapy must be kept constant for a period of at least 4 weeks prior to the Baseline Period
* Vagal nerve stimulation is allowed and will not be counted as a concomitant AED. The vagus nerve stimulation (VNS) device must be implanted for at least 6 months before Visit 1, and the device settings must be stable for at least 4 weeks before Visit 1 and be kept stable during the Baseline Period and the Treatment Period. Use of the VNS device magnet is allowed
* Body weight at Visit 1 is at least 4 kg for infants.
* Females of childbearing potential must have a negative pregnancy test at Visit 1
* Subjects with West Syndrome are eligible if Baseline EEG demonstrates hypsarrhythmia despite treatment with at least 2 AEDs appropriate for the treatment of this syndrome

Exclusion Criteria:

* Subject has previously participated in this study, subject has been assigned to Lacosamide (LCM) in a previous LCM study, or subject has ever received LCM
* Subject is currently participating or has participated within the last 2 months in any study of an investigational drug or experimental device
* Subject has a history of convulsive status epilepticus within 1 month prior to Visit 1
* Subject has a current or previous diagnosis of pseudoseizures, conversion disorders, or other nonepileptic ictal events that could be confused with seizures
* Subject has exclusively typical absence (Type IIA1) or atypical absence (Type IIA2) seizures (no other generalized seizure types are reported), or has only partial-onset seizures (Type I)
* Subject has any medical or psychiatric condition that, in the opinion of the investigator, could jeopardize the subject's health or would compromise the subject's ability to participate in this study
* Subject ≥6 years of age has a lifetime history of suicide attempt (including an actual attempt, interrupted attempt, or aborted attempt), or has suicidal ideation in the past 6 months as indicated by a positive response ("Yes") to either Question 4 or Question 5 of the Columbia Suicide Severity Rating Scale (C-SSRS) at Screening
* Subject has a known hypersensitivity to any components of the investigational medicinal product (IMP)
* Subject has a medical condition that could reasonably be expected to interfere with drug absorption, distribution, metabolism, or excretion
* Subject has a known history of severe anaphylactic reaction or serious blood dyscrasias
* Subject has any history of alcohol or drug abuse within the previous 2 years
* Subject has an acute or sub-acutely progressive central nervous system disease. Subject has epilepsy secondary to a progressing cerebral disease or any other progressively neurodegenerative disease (malignant brain tumor or Rasmussen Syndrome)
* Subject has alanine aminotransferase (ALT), aspartate aminotransferase (AST), or total bilirubin levels ≥2x the upper limit of normal (ULN) or has alkaline phosphatase levels ≥3x ULN
* Subject has impaired renal function (ie, creatinine clearance is lower than 30 mL/min) at Visit 1
* Subject has sick sinus syndrome without a pacemaker, or second or third degree atrioventricular (AV) block
* Subjects with second- or third-degree heart block are excluded from SP0966 (NCT01969851), without the requirement of being at rest
* Subject has hemodynamically significant heart disease (eg, heart failure)
* Subject has an arrhythmic heart condition requiring medical therapy
* Subject has a known cardiac sodium channelopathy, such as Brugada syndrome
* Female subject who is pregnant or nursing, and/or a female subject of childbearing potential who is not surgically sterile or does not practice 1 highly effective method of contraception (according to International Conference on Harmonisation [ICH] guidance. Female subject of childbearing potential taking enzyme inducing antiepileptic drugs(EI AEDs) (carbamazepine, phenytoin, barbiturates, primidone, topiramate, oxcarbazepine) who is not surgically sterile or does not practice 1 highly effective method of contraception according to the World Health Organization recommendation (ie, depot medroxyprogesterone acetate, norethisterone enantate, intrauterine devices, combined injectables, and progestogen implants) with administration of enzyme inducing antiepileptic drugs (EI-AEDs) or does not practice 2 combined methods of contraception (ie, combined hormonal contraception plus barrier method with spermicidal agent), unless sexually abstinent, for the duration of the study
* Subject has been treated with vigabatrin and experienced any vision loss. Subjects who have received vigabatrin in the past must have documentation of an assessment for vision loss prior to study entry or documentation of why visual field testing cannot be performed
* Subject has been treated with felbamate and has experienced any serious toxicity issues (defined as liver failure, aplastic anemia) with this treatment. Subjects treated with felbamate for less than 12 months are excluded. Note: any subject who has been treated with felbamate for at least 12 months and has not experienced serious toxicity issues is eligible
* Subject is taking monoamine oxidase (MAO) inhibitors or narcotic analgesics.
* Subject is on a ketogenic or other specialized diet. If he/she was on a specialized diet in the past, he/she must be off the diet for at least 2 months prior to the Screening Visit (Visit 1)
* Subject has primary generalized tonic-clonic seizures with a diagnosis of idiopathic generalized epilepsy

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 55 (Actual)
Dates: Start 2014-02-13 (Actual); Primary Completion 2018-04-10 (Actual); Study Completion 2018-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 844 599 2273
Locations (18):
- United States (6):
  - 103, Los Angeles, California
  - 101, Orlando, Florida
  - 104, Henderson, Nevada
  - 112, Hackensack, New Jersey
  - 108, New Brunswick, New Jersey
  - 107, Akron, Ohio
- France (2):
  - 309, Ile-De-France
  - 303, Lyon
- Hungary (5):
  - 701, Budapest
  - 702, Budapest
  - 703, Budapest
  - 704, Budapest
  - 705, Debrecen
- 154, Guadalajara, Mexico
- Poland (4):
  - 807, Katowice
  - 801, Krakow
  - 805, Lublin
  - 802, Szczecin

REFERENCES:
- [Derived] Auvin S, Arzimanoglou A, Beller C, Floricel F, Daniels T, Bozorg A. Safety, tolerability, and efficacy of adjunctive lacosamide in pediatric patients with epilepsy syndromes associated with generalized seizures: Phase 2, open-label exploratory trial. Epilepsia. 2023 Nov;64(11):2947-2957. doi: 10.1111/epi.17741. Epub 2023 Aug 23. PMID 37545406
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in February 2014 and concluded in April 2018.
Pre-assignment Details: The Participant Flow refers to the Safety Set which consisted of all enrolled subjects who took at least 1 dose of lacosamide (LCM).
Groups:
- Lacosamide 1 Month - <4 Years: Subjects, aged 1 month to <4 years, who were administered Lacosamide oral solution (for subjects weighing <50 kg) or tablet (for subjects weighing >=50 kg). The initial dose of 2 mg/kg/day (for subjects weighing <50 kg), or 100 mg/day (for subjects weighing >=50 kg) was titrated to optimize tolerability and seizure control to at least 4 mg/kg/day for subjects weighing <50 kg, or 200 mg/day for subjects weighing >=50 kg; not to exceed 12 mg/kg/day for subjects weighing <50 kg, or 600 mg/day in subjects weighing >=50 kg.
- Lacosamide 4 Years - <12 Years: Subjects, aged 4 years to <12 years, who were administered Lacosamide oral solution (for subjects weighing <50 kg) or tablet (for subjects weighing >=50 kg). The initial dose of 2 mg/kg/day (for subjects weighing <50 kg), or 100 mg/day (for subjects weighing >=50 kg) was titrated to optimize tolerability and seizure control to at least 4 mg/kg/day for subjects weighing <50kg, or 200 mg/day for subjects weighing >=50 kg; not to exceed 12 mg/kg/day for subjects weighing <50 kg, or 600 mg/day in subjects weighing >=50 kg.
- Lacosamide 12 Years - <18 Years: Subjects, aged 12 years to <18 years, who were administered Lacosamide oral solution (for subjects weighing <50 kg) or tablet (for subjects weighing >=50 kg). The initial dose of 2 mg/kg/day (for subjects weighing <50 kg), or 100 mg/day (for subjects weighing >=50 kg) was titrated to optimize tolerability and seizure control to at least 4 mg/kg/day for subjects weighing <50kg, or 200 mg/day for subjects weighing >=50 kg; not to exceed 12 mg/kg/day for subjects weighing <50 kg, or 600 mg/day in subjects weighing >=50 kg.
Period: Overall Study
Arm/Group | Lacosamide 1 Month - <4 Years | Lacosamide 4 Years - <12 Years | Lacosamide 12 Years - <18 Years
Started | 10 | 24 | 21
Completed | 9 | 21 | 14
Not Completed | 1 | 3 | 7
Not completed — Adverse Event | 0 | 0 | 3
Not completed — Lack of Efficacy | 0 | 3 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — No effective dose in Titration period | 0 | 0 | 1
Not completed — Sponsor decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Baseline Characteristics refer to the Safety Set which consisted of all enrolled subjects who took at least 1 dose of lacosamide (LCM).
Arm/Group | Lacosamide 1 Month - <4 Years | Lacosamide 4 Years - <12 Years | Lacosamide 12 Years - <18 Years | Total Title
Number analyzed (Participants) | 10 | 24 | 21 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 24 | 21 | 55
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.716 (0.765) | 6.969 (1.998) | 14.753 (1.766) | 9.168 (4.994)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 9 | 15 | 24
  Male | 10 | 15 | 6 | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 2
  Black or African American | 0 | 2 | 1 | 3
  White | 7 | 18 | 11 | 36
  More than one race | 3 | 3 | 7 | 13
  Unknown or Not Reported | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Changes in Count of Generalized Spike-wave Discharges on 24-hour Ambulatory Electroencephalogram (EEG) From Visit 2 to Visit 6
Description: The mean change in the count of generalized spike-wave discharges was presented. Visit 6 (Week 6) was the End of the Titration Period.
Time Frame: From Baseline (Day 1) to Visit 6 (Week 6)
Population: The Safety Set (SS) included all enrolled subjects who took at least 1 dose of lacosamide (LCM).
Measure: Mean (Standard Deviation); unit: discharges
Groups:
- Lacosamide 1 Month - <4 Years SS: Subjects, aged 1 month to <4 years, who were administered Lacosamide oral solution (for subjects weighing <50 kg) or tablet (for subjects weighing >=50 kg). The initial dose of 2 mg/kg/day (for subjects weighing <50 kg), or 100 mg/day (for subjects weighing >=50 kg) was titrated to optimize tolerability and seizure control to at least 4 mg/kg/day for subjects weighing <50 kg, or 200 mg/day for subjects weighing >=50 kg; not to exceed 12 mg/kg/day for subjects weighing <50 kg, or 600 mg/day in subjects weighing >=50 kg.
- Lacosamide 4 Years - <2 Years SS: Subjects, aged 4 years to <12 years, who were administered Lacosamide oral solution (for subjects weighing <50 kg) or tablet (for subjects weighing >=50 kg). The initial dose of 2 mg/kg/day (for subjects weighing <50 kg), or 100 mg/day (for subjects weighing >=50 kg) was titrated to optimize tolerability and seizure control to at least 4 mg/kg/day for subjects weighing <50kg, or 200 mg/day for subjects weighing >=50 kg; not to exceed 12 mg/kg/day for subjects weighing <50 kg, or 600 mg/day in subjects weighing >=50 kg.
- Lacosamide 12 Years - <18 Years SS: Subjects, aged 12 years to <18 years, who were administered Lacosamide oral solution (for subjects weighing <50 kg) or tablet (for subjects weighing >=50 kg). The initial dose of 2 mg/kg/day (for subjects weighing <50 kg), or 100 mg/day (for subjects weighing >=50 kg) was titrated to optimize tolerability and seizure control to at least 4 mg/kg/day for subjects weighing <50kg, or 200 mg/day for subjects weighing >=50 kg; not to exceed 12 mg/kg/day for subjects weighing <50 kg, or 600 mg/day in subjects weighing >=50 kg.
Arm/Group | Lacosamide 1 Month - <4 Years SS | Lacosamide 4 Years - <2 Years SS | Lacosamide 12 Years - <18 Years SS
Number analyzed (Participants) | 9 | 22 | 14
discharges | -4.55 (257.32) | -166.22 (447.80) | -203.12 (432.42)

2. Primary Outcome: Mean Change in Days With Any Generalized Seizures (Absence, Myoclonic, Clonic, Tonic, Tonic-clonic, Atonic, Partial Evolving to Secondarily Generalized) Per 28 Days From the Baseline Period to the Maintenance Period (Approximately 24 Weeks)
Description: The mean change in the count of days with generalized seizures was presented.
Time Frame: Baseline Period to the Maintenance Period (approximately 24 weeks)
Population: The Safety Set (SS) included all enrolled subjects who took at least 1 dose of lacosamide (LCM).
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Lacosamide 1 Month - <4 Years SS | Lacosamide 4 Years - <2 Years SS | Lacosamide 12 Years - <18 Years SS
Number analyzed (Participants) | 10 | 23 | 20
days | 0.50 (6.63) | -1.90 (3.76) | -3.38 (6.42)

3. Secondary Outcome: Mean Changes in Count of 3 Hz Spike-wave Discharges (During Waking Hours) on 24-hour Ambulatory EEG From Visit 2 to Visit 6
Description: The mean change in the count of 3 Hertz (Hz) spike-wave discharges was presented. Visit 6 (Week 6) was the End of the Titration Period.
Time Frame: From Baseline (Day 1) to Visit 6 (Week 6)
Population: The Safety Set (SS) included all enrolled subjects who took at least 1 dose of lacosamide (LCM).
Measure: Mean (Standard Deviation); unit: count of discharges
Arm/Group | Lacosamide 1 Month - <4 Years SS | Lacosamide 4 Years - <2 Years SS | Lacosamide 12 Years - <18 Years SS
Number analyzed (Participants) | 9 | 22 | 14
count of discharges | -0.14 (0.42) | -1.60 (9.92) | 0.00 (0.00)

4. Secondary Outcome: Number of Subject Withdrawals Due to Adverse Events From Baseline to End of Study (Approximately 32 Weeks)
Description: An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment.
Time Frame: From Baseline to End of Study (approximately 32 weeks)
Population: The Safety Set (SS) included all enrolled subjects who took at least 1 dose of lacosamide (LCM).
Measure: Count of Participants; unit: Participants
Arm/Group | Lacosamide 1 Month - <4 Years SS | Lacosamide 4 Years - <2 Years SS | Lacosamide 12 Years - <18 Years SS
Number analyzed (Participants) | 10 | 24 | 21
Participants | 0 | 0 | 3

5. Secondary Outcome: Number of Subjects Experiencing at Least 1 Treatment-emergent Adverse Event From Baseline to End of Study (Approximately 32 Weeks)
Description: as for outcome 4
Time Frame: From Baseline to End of Study (approximately 32 weeks)
Population: The Safety Set (SS) included all enrolled subjects who took at least 1 dose of lacosamide (LCM).
Measure: Count of Participants; unit: Participants
Arm/Group | Lacosamide 1 Month - <4 Years SS | Lacosamide 4 Years - <2 Years SS | Lacosamide 12 Years - <18 Years SS
Number analyzed (Participants) | 10 | 24 | 21
Participants | 10 | 21 | 18

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the study (up to week 26)
Description: An Adverse Event (AE) was any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product that did not necessarily have a causal relationship with this treatment.
Arm/Group | Lacosamide 1 Month - <4 Years | Lacosamide 4 Years - <12 Years | Lacosamide 12 Years - <18 Years
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/24 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/24 | 1/21
Other Adverse Events (participants affected / at risk) | 10/10 | 19/24 | 15/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide 1 Month - <4 Years (N=10) | Lacosamide 4 Years - <12 Years (N=24) | Lacosamide 12 Years - <18 Years (N=21)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide 1 Month - <4 Years (N=10) | Lacosamide 4 Years - <12 Years (N=24) | Lacosamide 12 Years - <18 Years (N=21)
Vomiting (Gastrointestinal disorders) | 0 (0) | 4 (5) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 4 (5) | 6 (7) | 3 (3)
Irritability (General disorders) | 1 (1) | 1 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 5 (7) | 1 (1) | 3 (3)
Pharyngotonsillitis (Infections and infestations) | 2 (2) | 1 (2) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 4 (4) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2) | 2 (3)
Pharyngitis (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
Ear infection (Infections and infestations) | 1 (3) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2)
Somnolence (Nervous system disorders) | 4 (4) | 2 (2) | 2 (3)
Headache (Nervous system disorders) | 1 (6) | 0 (0) | 4 (7)
Tremor (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-03-06): https://cdn.clinicaltrials.gov/large-docs/51/NCT01969851/SAP_000.pdf
  • Study Protocol (2015-02-26): https://cdn.clinicaltrials.gov/large-docs/51/NCT01969851/Prot_001.pdf